CLINICAL TRIAL: NCT05909150
Title: Use of Hypertonic Saline Solution to Prevent Acute Kidney Injury After Heart Transplantation
Brief Title: Hypertonic Saline Solution to Prevent Acute Kidney Injury After Heart Transplantation
Acronym: HSS-HT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fernando Bacal (Other)
Responsible Party: Sponsor-Investigator, Fernando Bacal, Director of Heart Transplant Unit (Heart Institute)., University of Sao Paulo General Hospital
Organization: University of Sao Paulo General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSS-HT
Record Dates: First submitted 2023-03-24; First posted 2023-06-18 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Heart Transplantation; Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hypertonic Saline Solution 3,5% (HSS) (Active Comparator)
  Interventions: Drug: Sodium chloride solution 3,5%
- Normal Saline Solution (NS) (Placebo Comparator)
  Interventions: Drug: Sodium chloride solution 0,9%

INTERVENTIONS:
Drug: Sodium chloride solution 3,5% — Patients will receive 150 mL HSS 3,5% intravenous twice daily for 3 days after heart transplantation.
  Arms: Hypertonic Saline Solution 3,5% (HSS)
Drug: Sodium chloride solution 0,9% — Patients will receive 150 mL NS 0,9% intravenous twice daily for 3 days after heart transplantation.
  Arms: Normal Saline Solution (NS)

SUMMARY:
The goal of this study is to evaluate if hypertonic saline solution can prevent or attenuate acute kidney injury after heart transplantation in the early postoperative phase.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a frequent complication immediately after heart transplantation (HT), with incidence rates between 40-70%. Several factors contribute to this complication, such as hypervolemia, hyperactivation of renin-angiotensin-aldosterone system (RASS) and low cardiac output. Hypertonic saline solution (HSS) can reduce diuretic resistance, increase urinary output and improve renal function in hypervolemic status such as acute heart failure. Therefore, the investigators hypothesized that the use of HSS could prevent or attenuate AKI after heart transplantation in the early postoperative phase. The investigators aim to randomize 74 patients to receive 150 mL of HSS 3,5% or placebo (saline solution 0,9%) twice daily for 3 days after HT. Renal function, right ventricular echocardiographic parameters and pulmonary artery catheter parameters will be assessed. Patients will be followed-up until 30 days, or death.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients submitted to orthotopic heart transplantation (HT)

Exclusion Criteria:

* Requirement of renal replacement therapy at the time of HT
* Requirement of extracorporeal membrane oxygenation (ECMO) before or immediately after HT
* Severe peri-operative mechanical complications
* Double transplant (e.g. heart-kidney or heart-lung)
* Hypernatremia (Na ≥ 145)
* Severe hyponatremia (Na ≤ 120)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Prevention of acute kidney injury | Days 3 -7 post-transplantation
  Demonstrate a peak value of creatinine 30% lower in the active arm

SECONDARY OUTCOMES:
Mortality | 30 days
  Incidence of all cause mortality during the first 30 days after start of the study
Incidence of acute kidney injury requiring hemodialysis | 30 days
  Rate of patients which required hemodialysis during the first 30 days after start of the study
Intensive care unit (ICU) length of stay | During ICU stay, an average of 5 days
  The time frame between start of the study and ICU discharge will be calculated.
Time to wean inotropes and vasopressors | During ICU stay, an average of 5 days
  Time to wean all inotropes and vasopressors will be calculated.
Incidence of right ventricular dysfunction | Until day 5 post-transplantation
  Right ventricular dysfunction will be assessed through the following echocardiographic parameters:
  * Tricuspid annular plane systolic excursion (TAPSE; normal ≥1.7 cm);
  * Tricuspid annular velocity (S') (normal ≥9.5 cm/s);
  * Fractional area change (FAC; normal ≥35 percent);
  * Right Ventricle basal diameter (normal ≤4.1 cm)
Hypertonic saline solution (HSS) hemodynamic effect | Until day 3 post-transplantation
  Pulmonary artery catheter measures will be assessed before HSS infusion, immediately after HSS infusion and 30 min after HSS infusion.
  The following measures will be assessed:
  * Right atrial pressure (RAP)
  * Systolic pulmonary artery pressure (sPAP)
  * Diastolic pulmonary artery pressure (dPAP)
  * Mean pulmonary artery pressure (mPAP)
  * Pulmonary artery wedge pressure (PCWP)
  * Cardiac output (CO)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Bacal, PhD, Study Director — University of Sao Paulo
Locations (1):
- Heart Institute, University of São Paulo., São Paulo, Brazil